CLINICAL TRIAL: NCT01385202
Title: THERMOCOOL® SMARTTOUCH™ Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Smart-AF
Record Dates: First submitted 2011-06-27; First posted 2011-06-30 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Heart Diseases; Arrhythmia; Atrial Fibrillation
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac; Atrial Fibrillation

ARMS (1):
- THERMOCOOL® SMARTTOUCH™ Catheter (Experimental)
  Interventions: Device: THERMOCOOL® SMARTTOUCH™ Catheter

INTERVENTIONS:
Device: THERMOCOOL® SMARTTOUCH™ Catheter — AF Ablation

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the THERMOCOOL® SMARTTOUCH™ Catheters with Contact Force Sensing Capability in the treatment of drug refractory symptomatic paroxysmal Atrial Fibrillation (AF) during standard electrophysiology mapping and RF procedures.

ELIGIBILITY:
Inclusion Criteria:

* Have had at least 3 atrial fibrillation episodes within 6 months of this study
* Have failed at least one antiarrhythmic drug shown by repeated atrial fibrillation episodes
* 18 years of age or older

Exclusion Criteria:

* Have had previous ablation for atrial fibrillation
* Have take amiodarone within 6 months of this study
* Have had any heart surgery within the last 60 days
* Have had a heart attack within the last 60 days
* Females who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Study Chair — Texas Cardiac Arrhythmia Research; David J Wilber, MD, Study Chair — Loyola University; Francis E Marchlinski, MD, Study Chair — University of Pennsylvania; Douglas L Packer, MD, Study Chair — Mayo Clinic; Hiroshi Nakagawa, MD, Ph.D., Study Chair — University of Oklahoma; Hans Kottkamp, MD, Study Chair — University Leipzig

REFERENCES:
- [Derived] Reddy VY, Pollak S, Lindsay BD, McElderry HT, Natale A, Kantipudi C, Mansour M, Melby DP, Lakkireddy D, Levy T, Izraeli D, Sangli C, Wilber D. Relationship Between Catheter Stability and 12-Month Success After Pulmonary Vein Isolation: A Subanalysis of the SMART-AF Trial. JACC Clin Electrophysiol. 2016 Nov;2(6):691-699. doi: 10.1016/j.jacep.2016.07.014. Epub 2016 Nov 21. PMID 29759747
- [Derived] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on June 02, 2011. Twenty-one (21) sites enrolled subjects. Last patient enrolled on December 22, 2011. Last procedure on December 29, 2011.
Groups:
- THERMOCOOL® SMARTTOUCH™ Catheter: THERMOCOOL® SMARTTOUCH™ Deflectable Diagnostic/Ablation Catheter
Period: Overall Study
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Started | 172 (Per protocol, enrolled subjects were defined as those who signed inform consent form.)
Study Catheter Inserted | 161
Undergoing Ablation | 160
Completed | 154
Not Completed | 18
Not completed — Lost to Follow-up | 6
Not completed — Not Eligible | 11
Not completed — Withdrawn | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects, including all who signed inform consent form.
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 168
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 165
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 172

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Subjects Who Were Free From Documented Symptomatic Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atrial Flutter (AFL) Episodes Through 12-month Follow-up
Description: The primary effectiveness endpoint for this study will be freedom from documented symptomatic atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) episodes through 12-month follow-up (includes a three month blanking period).
Time Frame: 12-months
Population: Primary Effectiveness Cohort includes those enrolled who met the inclusion/exclusion criteria and had undergone insertion of the study catheter and Atrial Fibrillation (AF) ablation procedure, excluding those with radiofrequency energy not delivered, with calibration roll-in, and with only non-study arrhythmia.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 114
percentage of participants | 70.2 [60.9 to 78.4]
Statistical Analysis 1: Comparison: THERMOCOOL® SMARTTOUCH™ Catheter; The null hypothesis was that the rate of freedom from documented symptomatic AF/AFL/AT at 12 months would be less than or equal to the pre-determined performance criterion of 50%. The alternative hypothesis was that the rate of freedom from documented symptomatic AF/AFL/AT at 12 months would be greater than the pre-determined performance criterion of 50%; Test type: Superiority or Other; p < 0.0001, Fisher Exact — In the worst-case scenario analysis, over seventy-percent (70.2%, 80/114) of the primary effectiveness cohort (PEC) were free from documented symptomatic atrial tachyarrhythmias during their effectiveness evaluation period; The lower bound of the 95% confidence intervals was 60.9%, significantly higher than the pre-determined performance goal of 50% (p<0.0001); Primary effectiveness rate = 70.2, 95% CI 2-sided [60.9 to 78.4] — The confidence intervals above are the 95% exact binomial confidence intervals
Statistical Analysis 2: Comparison: THERMOCOOL® SMARTTOUCH™ Catheter; Test type: Superiority or Other; Primary effectiveness rate = 74, 95% CI 2-sided [66 to 82] — The 95% confidence intervals above were calculated using the Kaplan-Meier (KM) method

2. Primary Outcome: Incidence of Early Onset (Within 7 Days of the AF Ablation Procedure) Primary Adverse Events.
Description: Primary adverse events (AE) include Death, Myocardial infarction (MI), Pulmonary vein (PV) stenosis, Diaphragmatic paralysis, Atrio-esophageal fistula, Transient Ischemic Attack (TIA), Stroke / Cerebrovascular accident (CVA), Thromboembolism, Pericarditis, Cardiac Tamponade, Pericardial effusion, Pneumothorax, Atrial perforation, Vascular Access Complications, Pulmonary edema, Hospitalization (initial and prolonged), and Heart block.
Time Frame: 7 days of the AF ablation procedure
Population: Safety cohort includes all enrolled subjects who had the study catheter inserted.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with primary AE
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Number analyzed (Participants) | 161
Percentage of patients with primary AE | 9.9 [5.8 to 15.6]

3. Secondary Outcome: Rate of Acute Success
Description: Acute success is defined as confirmation of entrance block in all Pulmonary veins (PV).
Time Frame: End of procedure
Population: The analysis population for this endpoint includes two groups; a): Calibration Roll-in subjects who were prospectively identified prior to the study procedure and b) the Effectiveness Cohort. Both groups underwent an AF ablation procedure with the study catheter.
Measure: Number; unit: percentage of participants
Groups:
- THERMOCOOL® SMARTTOUCH™ Catheter-Effective Cohort: THERMOCOOL® SMARTTOUCH™ Deflectable Diagnostic/Ablation Catheter.
- Calibration Roll-in: Calibration roll-in case(s) is intended to calibrate an investigator's tactile feel, catheter manipulation technique, and use of other surrogate measures (electrogram signal, impedance, etc.) during the procedure.
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter-Effective Cohort | Calibration Roll-in
Number analyzed (Participants) | 122 | 38
percentage of participants | 100 | 94.7

ADVERSE EVENTS:
Arm/Group | THERMOCOOL® SMARTTOUCH™ Catheter
Serious Adverse Events (participants affected / at risk) | 38/161
Other Adverse Events (participants affected / at risk) | 70/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL® SMARTTOUCH™ Catheter (N=161)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 4 (5)
HEART BLOCK (Cardiac disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Cardiac disorders) | 12 (17)
PAF ABLATION REDO (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 3 (3)
VASOVAGAL SYNCOPE BECAUSE OF LEG CRAMPS (Cardiac disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Gastrointestinal disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
VIRAL INFECTION RESULTING IN HOSPITALIZATION, PHLEBITIS FROM IV (Infections and infestations) | 1 (1)
WBC ELEVATED, ABDOMINAL PAIN, ILEUS AND LOSS OF CAPTURE IN RV LEAD POST-LASER LEAD EXTRACT (Infections and infestations) | 1 (1)
CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Musculoskeletal and connective tissue disorders) | 2 (2)
LEFT KNEE INJURY (Musculoskeletal and connective tissue disorders) | 1 (1)
LEFT ARM PAIN (Nervous system disorders) | 1 (1)
LOC (Nervous system disorders) | 1 (1)
MIGRAINES (Nervous system disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Renal and urinary disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Respiratory, thoracic and mediastinal disorders) | 2 (2)
LUNG MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Vascular disorders) | 4 (4)
VASCULAR ACCESS COMPLICATIONS (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL® SMARTTOUCH™ Catheter (N=161)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
AF (Cardiac disorders) | 1 (1)
AFLUTTER (Cardiac disorders) | 1 (1)
AORTIC ROOT DILATION (Cardiac disorders) | 1 (1)
ARRHYTHMIA -FLUTTER (Cardiac disorders) | 1 (1)
ARRYTHMIA (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION RECURRENCE (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION, FLUTTER (Cardiac disorders) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 2 (3)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1)
BILATERAL LOWER EXTREMITY EDEMA AND PAIN (Cardiac disorders) | 1 (1)
BREAKTHROUGH A-FIB (Cardiac disorders) | 1 (1)
CARDIOVERSION FOR ATRIAL TACH (Cardiac disorders) | 1 (1)
CHEST DISCOMFORT (Cardiac disorders) | 1 (1)
EXERTIONAL ANGINA (Cardiac disorders) | 1 (1)
HEART RACING, LIGHTHEADED, CHEST PAIN (Cardiac disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Cardiac disorders) | 2 (2)
HYPOTENSION (Cardiac disorders) | 2 (2)
NEAR-SYNCOPAL EPISODES (Cardiac disorders) | 1 (1)
NEW DIAGNOSIS OF ATYPICAL ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 2 (2)
PERICARDITIS (Cardiac disorders) | 2 (2)
PERICARDIUM STAIN (Cardiac disorders) | 1 (1)
RAPID ATRIAL FIB (Cardiac disorders) | 1 (1)
RAPID ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
RECURRENCE AFIB REQUIRING CVS (Cardiac disorders) | 1 (1)
RECURRENCE OF AF REQUIRING CARDIOVERSION (Cardiac disorders) | 2 (2)
RECURRENCE OF AFIB REQUIRING REPEAT ABLATION (Cardiac disorders) | 1 (1)
RECURRENT AF REQUIRING CARDIOVERSION (Cardiac disorders) | 1 (1)
REPEAT PULMONARY VEIN ISOLATION (Cardiac disorders) | 1 (1)
RIGHT SIDED ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
STRONG HEART BEAT (Cardiac disorders) | 1 (1)
VASOVAGAL EVENT (Cardiac disorders) | 1 (1)
VOLUME OVERLOAD (Cardiac disorders) | 1 (1)
ADRENAL GLAND MASS (Endocrine disorders) | 1 (1)
BLURRED VISION (Eye disorders) | 1 (1)
BLURRY VISION, TINNITUS, HEADACHE (Eye disorders) | 1 (1)
CHEST PAIN (Gastrointestinal disorders) | 1 (1)
DIAHRRHEA / STOMACH VIRUS (Gastrointestinal disorders) | 1 (1)
DIARRHEA , GAS (Gastrointestinal disorders) | 1 (1)
GERD, TROUBLE SWALLOWING (Gastrointestinal disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Gastrointestinal disorders) | 2 (2)
INTERMITTENT GASTRIC BURNING (Gastrointestinal disorders) | 1 (1)
NEW ONSET DIABETES (Gastrointestinal disorders) | 1 (1)
STOMACH VIRUS (Gastrointestinal disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
INCREASED TEMPERATURE (General disorders) | 1 (1)
WASHED OUT FEELING (General disorders) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Infections and infestations) | 1 (1)
SINUS INFECTION (Infections and infestations) | 2 (3)
SINUSITIS/BRONCHITIS (Infections and infestations) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 2 (2)
FALL - DUE TO SLIP (Injury, poisoning and procedural complications) | 1 (1)
ADHESIVE CAPSULITIS OF SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BRONCHITIS (Musculoskeletal and connective tissue disorders) | 2 (2)
CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
EAR INFECTION (Musculoskeletal and connective tissue disorders) | 1 (1)
HOSPITALIZATION, INTIAL AND PROLONGED (Musculoskeletal and connective tissue disorders) | 1 (1)
LEFT SHOULDER/ARM PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PARTIAL KNEE REPLACEMENT (Musculoskeletal and connective tissue disorders) | 1 (1)
PINCHED NERVES (Musculoskeletal and connective tissue disorders) | 1 (1)
PLANTER FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
REPAIR OF BICEP TENDON (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNOVIAL OSTEOCHONDROMATOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
UPPER SHOULDER/CERVICAL SPINE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BENIGN TUMOR FOUND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
HEADACHE WITH BLURRED VISION (Nervous system disorders) | 1 (1)
MIGRAINE HEADACHE WITH VISUAL FIELD LOSS (Nervous system disorders) | 1 (1)
MIGRANE HEADACHE (Nervous system disorders) | 1 (1)
PAIN, NUMBNESS -LEFT HAND/FINGERS LOSS OF STRENGTH (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
VASCULAR ACCESS COMPLICATIONS (Nervous system disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ONGOING EXERTIONAL SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 4 (4)
SOB AND BLOOD TRANSFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BLEEDING GUMS (Vascular disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 2 (2)
POSSIBLE HEMATOMA (Vascular disorders) | 1 (1)
RECTAL BLEEDING (Vascular disorders) | 1 (1)
RIGHT GROIN HEMATOMA (Vascular disorders) | 1 (1)
RT GROIN SEROMA/HEMATOMA (Vascular disorders) | 1 (1)
SIDE EFFECTS FROM MEDICATION DOSING (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.